CLINICAL TRIAL: NCT02720627
Title: An Open Label Evaluation of the Adrenal Suppression Potential and Trough Plasma Concentrations of Cortexolone 17α-Propionate (CB-03-01) Cream Applied Every 12 Hours for Two Weeks in Subjects 9 to <12 Years of Age With Acne Vulgaris
Brief Title: An Evaluation of the Adrenal Suppression Potential and PK of CB-03-01 Cream in Pediatric Patients With Acne Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cassiopea SpA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CB-03-01/28
Record Dates: First submitted 2016-03-22; First posted 2016-03-28 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Acne Vulgaris
Keywords: acne; cortexolone; anti-androgen
MeSH Terms: conditions — Acne Vulgaris | interventions — Clascoterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CB-03-01 cream, 1% (Experimental): Topical CB-03-01 (cortexolone 17α-propionate) cream containing 1% active drug applied to the face and trunk twice daily for 14 days
  Interventions: Drug: cortexolone 17α-propionate

INTERVENTIONS:
Drug: cortexolone 17α-propionate — CB-03-01 cream is a topical steroidal antiandrogen that is being developed for the potential treatment of acne vulgaris, an androgen-dependent skin disorder.
  Other Names: CB-03-01

SUMMARY:
This study is designed to determine the hypothalamic-pituitary-adrenal (HPA) axis suppression potential and pharmacokinetic (PK) properties of CB-03-01 Cream, 1%, applied every twelve hours for two weeks, in pediatric patients 9 to less than 12 years of age with acne vulgaris. Adrenal suppression effects and systemic safety are an important safety concern. The current study is designed to investigate these potential concerns under maximal use conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patient must provide written informed assent and be accompanied by the parent or legal guardian at the time of assent/consent signing. The parent or legal guardian must provide written informed consent for the patient.
* Patient has moderate to severe facial acne vulgaris as determined by the Investigator and obvious acne on the trunk (i.e., shoulders, upper chest, and/or back).
* Females of childbearing potential must be using highly effective birth control methods with a negative urine pregnancy test (UPT) at study start.
* Patient must be in general good health with normal renal function and no clinically relevant abnormalities present at study start.
* Patient and parent/guardian are able to communicate with the staff and are willing to comply with study instructions, reside at and/or return to the clinic for required visits.

Exclusion Criteria:

* Patient is pregnant, lactating, or is planning to become pregnant during the study.
* Patient has a Body Mass Index (BMI) for age percentile > 95%.
* Patient has any skin or medical condition, including facial hair that could interfere with the evaluation of the test article or requires the use of interfering topical or systemic therapy.
* Patient has received an investigational drug or been treated with an investigational device within 30 days prior to study start.
* Patient is currently enrolled in an investigational drug or device study.
* Patient has any condition which, in the investigator's opinion, would make it unsafe for the patient to participate in this research study.
* Patient has known allergy or sensitivity to CB-03-01 or any of its ingredients
* Patient has participated in a previous CB-03-01 study.

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2016-10-28 (Actual); Primary Completion 2018-03-21 (Actual); Study Completion 2018-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R&D Department, Study Director — Cassiopea SpA
Locations (10):
- United States (3):
  - Site 103, Fort Smith, Arkansas
  - Site 101, San Diego, California
  - Site 102, Houston, Texas
- Poland (7):
  - Site 4814, Częstochowa
  - Site 4811, Katowice
  - Site 4813, Krakow
  - Site 4815, Krakow
  - Site 4816, Rzeszów
  - Site 4812, Szczecin
  - Site 4817, Tarnów

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- CB-03-01 Cream, 1%: Topical CB-03-01 (cortexolone 17α-propionate) cream containing 1% active drug applied to the face and trunk twice daily for 14 days
  cortexolone 17α-propionate (USAN/INN: clascoterone): is a topical steroidal antiandrogen that is being developed for the potential treatment of acne vulgaris, an androgen-dependent skin disorder.
Period: Overall Study
Arm/Group | CB-03-01 Cream, 1%
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety Population, defined as all enrolled subjects who were dispensed and applied at least one dose of the test article. All enrolled subjects were included in the safety population.
Arm/Group | CB-03-01 Cream, 1%
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.2 (0.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0
Baseline HPA Axis Response [Mean (Standard Deviation); unit: mcg/dL] — Measurement of serum cortisol concentrations after stimulation of the adrenal cortex with cosyntropin (Cosyntropin Stimulation Test - CST). Hypothalamic-pituitary-adrenal (HPA) axis suppression is defined as a post-stimulation serum cortisol level ≤ 18 μg/dL at Day 14. Population: Evaluable Population, defined as all subjects in the Safety population who had evaluable cortisol assay data.
  mcg/dL
    Cortisol Level (Pre-CST): number analyzed (Participants) | 23
    Cortisol Level (Pre-CST) | 13.53 (4.53)
    Cortisol Level (Post-CST): number analyzed (Participants) | 23
    Cortisol Level (Post-CST) | 24.87 (3.70)

OUTCOME MEASURES:

1. Primary Outcome: Change in HPA Axis Response as Measured by CST
Description: Measurement of serum cortisol concentrations after stimulation of the adrenal cortex with cosyntropin (Cosyntropin Stimulation Test - CST). HPA axis suppression is defined as a post-stimulation serum cortisol level ≤ 18 μg/dL at Day 14.
Time Frame: Pre- and Post-CST on Day 14
Population: Evaluable population, defined as all subjects in the safety population who had evaluable cortisol assay data.
Measure: Mean (Standard Deviation); unit: mcg/dL
Arm/Group | CB-03-01 Cream, 1%
Number analyzed (Participants) | 23
mcg/dL
  Cortisol level (Pre-CST) | 12.50 (4.90)
  Cortisol level (Post-CST) | 22.95 (3.20)

2. Secondary Outcome: Evaluate Trough Plasma Concentrations
Description: Trough (single blood draw approximately 12 hours post the most recent dose) measurements of cortexolone 17α-propionate (clascoterone) concentration in plasma at Screening, Baseline, Day 7 and Day 14.
Time Frame: 14 Days
Population: The pharmacokinetic (PK) population included those subjects in the Safety population who had at least an 80% dose compliance based on number of applications, had at least one post-baseline PK blood draw within ±2 days of the scheduled visit at Days 7 and 14, and did not have any significant protocol deviations.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CB-03-01 Cream, 1%
Number analyzed (Participants) | 25
ng/mL
  Screening | 0.0 (0.0)
  Baseline (Day 1) | 0.027 (0.136)
  Day 7 | 0.577 (1.01)
  Day 14 | 0.606 (0.701)

ADVERSE EVENTS:
Time Frame: 14 Days or up to 42 days for those with laboratory evidence of adrenal suppression (i.e., post-stimulation serum cortisol level ≤18 μg/dL at Day 14).
Description: Any treatment emergent AEs ongoing at the end of the treatment period (Day 14) were followed until they resolve, the condition stabilizes, the events are otherwise explained, or the subject is lost to follow-up. In addition, all SAEs were followed until resolution as previously stated for study product-related AEs. Subjects with laboratory evidence of adrenal suppression at Day 14 were required to be re-tested 4 weeks later (Day 42); all four subjects returned to normal HPA function.
Groups:
- CB-03-01 Cream, 1%: Topical CB-03-01 (cortexolone 17α-propionate) cream containing 1% active drug applied to the face and trunk twice daily for 14 days
  cortexolone 17α-propionate (USAN/INN: clasocoterone): is a topical steroidal antiandrogen that is being developed for the potential treatment of acne vulgaris, an androgen-dependent skin disorder.
Arm/Group | CB-03-01 Cream, 1%
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 5/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CB-03-01 Cream, 1% (N=27)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
ACTH stimulation test abnormal (Investigations) | 4 (4) — Adrenocorticotropic Hormone (ACTH) stimulation testing is conducted by the Cosyntropin Stimulation Test.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor has first right to publish pooled study data. In the event that such manuscript has not been submitted for publication within 18 months from study completion/termination at all participating sites, the PI shall have the right to single center publications provided they submit any data for presentation, oral or written, to the Sponsor for review 60 days prior to public disclosure. The PI may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2016-02-18): https://cdn.clinicaltrials.gov/large-docs/27/NCT02720627/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-17): https://cdn.clinicaltrials.gov/large-docs/27/NCT02720627/SAP_001.pdf